CLINICAL TRIAL: NCT01769131
Title: A Comparison of Two Instruments for Stabilization of the Cervix During Office Procedures
Acronym: OB39
Status: Completed | Type: Observational
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Isaiah Johnson, Physician, Carilion Clinic
Other Study IDs: OB39
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Comparing Two Clamps for Mobilization of the Cervix During Common Gynecologic Office Procedures
Keywords: cervix; Allis; Tenaculum; gynecology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Allis
- Tenaculum

SUMMARY:
An Allis clamp causes less pain and bleeding than a single tooth tenaculum when used for mobilization of the cervix during common gynecologic office procedures.

The primary object is to determine the presence of a difference in pain perception between the two instruments.

The secondary objective is to evaluate the differences in the frequency of bleeding, that requires treatment, after removal of the instrument and the need to use an alternative instruments.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18 and 89 years of age
* Undergoing an IUD placement

Exclusion Criteria:

* IUD placement within the last 6 months
* Active cervical or pelvic infection
* pregnant
* Patient taking coagulation medications

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females between the ages of 18 and 89 years undergoing an IUD placement
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
A comparison of two instruments for stabilization of the cervix during office procedures | 1 year
  Primary - to determine the presence of a difference in pain perception between the two instruments.

SECONDARY OUTCOMES:
A comparison of two instruments for stabilization of the cervix during office procedures | 1 year
  Secondary - To evaluate the differences in the frequency of bleeding, that required treatment, after removal of the instruct and the need to use an alternative instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States